CLINICAL TRIAL: NCT05690282
Title: Randomized Controlled Trial Comparing Multimodal Pain Protocol Versus Hydrocodone-Acetaminophen for Post-Operative Pain Management in Orthopaedic Surgery Patients
Brief Title: Comparing Perioperative Outcomes in Pain Control
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, William Kent, Assistant Professor of Orthopaedic Surgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210031
Record Dates: First submitted 2022-12-19; First posted 2023-01-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard oral hydrocodone-acetaminophen post-op management (No Intervention)
- Multimodal pain post-op management (Ibuprofen/Acetaminophen/GABAPentin/0.25%Bupivacaine) (Active Comparator)
  Interventions: Drug: Multimodal Pain Management (Ibuprofen/Acetaminophen/GABAPentin/0.25%Bupivacaine)

INTERVENTIONS:
Drug: Multimodal Pain Management (Ibuprofen/Acetaminophen/GABAPentin/0.25%Bupivacaine) — Multimodal Pain Management to minimize patients' reliance on opioids.
  Arms: Multimodal pain post-op management (Ibuprofen/Acetaminophen/GABAPentin/0.25%Bupivacaine)

SUMMARY:
This project consists of a randomized controlled study design. Study candidates will include all patients 18 years or older, who were evaluated at UCSD and found to have an orthopaedic injury requiring surgery. Patients who consent to study participation will be randomized to receive either the multimodal pain management protocol or standard oral hydrocodone-acetaminophen for post-operative pain management. Data on opioid usage, pain control, and functional status will be collected for each participant. After 3 years of data collection, investigators will analyze this data to provide further insight in determining appropriateness of pain regimens that reduce the overall opioid consumption. Given the widespread opioid epidemic, it is imperative to develop alternative means to appropriately manage pain in orthopaedic surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic injury requiring surgery
* Evaluation and treatment at UCSD
* Age 18years or older
* Ability to understand the content of the patient information/Informed Consent Form
* Signed and dated Institutional Review Board (IRB) approved written informed consent

Exclusion Criteria:

* Polytrauma
* Any not medically managed severe systemic disease
* Their doctor has decided that it is in the patient's best interest to receive pain management regimen of one type vs. the other.
* The patient prefers one type of pain management protocol and is not willing to be randomized.
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment or confound pain control
* Pregnancy or women planning to conceive within the subject participation period (1 year)

  o Pregnancy will be self-reported and no test will be performed to test for it.
* Prisoner
* Participation in any other pharmacologic or medicinal product study within the previous month that could influence the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Morphine equivalents used | 1 year
  Morphine equivalents used over 1 year

SECONDARY OUTCOMES:
Pain Score (0-10, 0=no pain, 10=most severe pain) | 1 year
Number of Complications | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No